CLINICAL TRIAL: NCT04620928
Title: Defining the Neural Dynamics of Concept Retrieval Using Electrocorticography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, William L Gross, MD PhD, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO00038561
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: Present a behavioral intervention to a single group of participants and measure subsequent electrical activity in the brain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concept Retrieval (Experimental): Patients will be given behavioral intervention, and their brain activity recorded.
  Interventions: Behavioral: Concepts

INTERVENTIONS:
Behavioral: Concepts — Images and sounds that are characteristic of various common objects.

SUMMARY:
This study will look at the way activity within the brain changes over time while a person is trying to think about certain everyday concepts. To measure brain activity accurately, we will be using electrodes placed on people's brains during awake brain surgery.

DETAILED DESCRIPTION:
This study will measure the dynamics of cortical activity among early modal cortex and multimodal cortical regions during conceptual retrieval using electrocorticography. Participants will be patients undergoing awake temporal lobe craniotomies. During the surgery patients will have multiple high-density grids placed to simultaneously record activity in multiple areas while the patient is performing language tasks. Activity in each of these regions will be tested for timing differences and informational directionality to determine the temporal dynamics.

ELIGIBILITY:
Inclusion Criteria:

* Clinically determined to require an awake left temporal resection of a brain lesion with concurrent language testing.
* English as a first language.

Exclusion Criteria:

* Significant preoperative neuropsychological deficits in memory or naming.
* Patients with inability to make decisions regarding their participation in this research project.
* Surgeon does not plan to expose the area of interest or determines that recording during the resection will interfere with his surgical plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Brain activity | Recorded immediately during experiment
  Electrocorticographic brain activity measured from brain surface

CONTACTS AND LOCATIONS:
Overall Officials: William Gross, MD, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No